CLINICAL TRIAL: NCT02201888
Title: Effects of a Cognitive Rehabilitation Program: a Neurocognitive Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salvador Sarró, MD (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Centro de Investigación Biomédica en Red de Salud Mental (Network); Hermanas Hospitalarias del Sagrado Corazón de Jesús, Spain (Unknown)
Responsible Party: Sponsor-Investigator, Salvador Sarró, MD, Chief administrator, FIDMAG Germanes Hospitalàries
Organization: FIDMAG Germanes Hospitalàries (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-2009-15; PI09/90483 (Other: Instituto de Salud Carlos III)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Rehabilitation; Cognition
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Computer-assisted cognitive training (Experimental): Patients in this arm of the trial carried out computerized online training drawn from the Feskits program (www.feskits.com), chosen to have attention, memory and executive function components. Specifically the sessions included the following exercises: sustained attention (4 minutes), attention/perception (5 minutes), working memory (8 minutes), auditory and visual memory (8 minutes), executive function (10 minutes), language (6 minutes), and games (4 minutes).
  Interventions: Behavioral: Computer-assisted cognitive training
- Computerized active condition (Active Comparator): Patients allocated to this condition completed the same number of sessions as the cognitive training group but followed a computerized typing program (www.rapidtyping.com). This had similar design characteristics to the CRT condition, in that it was hierarchically organized with exercise level of difficulty being adjusted to the individual's level of performance and feedback being given at the end of each exercise. Additionally, patients in this condition played computerized games requiring typing (crosswords, word puzzles, etc) and were taught basic internet navigation by a supervisor. Exposure to the computer was of equivalent duration to the CRT condition.
  Interventions: Other: Computerized active condition
- Treatment as usual (Placebo Comparator): Patients in this condition participated in their (individually variable) daily rehabilitative activities. Patients allocated to the other two conditions also participated in these activities
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Computer-assisted cognitive training — Treatment lasted six months. The CRT and CC conditions consisted of biweekly sessions of 45 minutes. Patients in both conditions trained in groups of up to 8, supervised by a single person. The CRT and CC groups were scheduled at different times. The same personnel supervised both treatment conditions. All supervisors were trained by the coordinator of the study in the technical management of the two conditions.
  Other Names: Computer-assisted cognitive training (CRT)
  Arms: Computer-assisted cognitive training
Other: Computerized active condition — Treatment lasted six months. The CRT and CC conditions consisted of biweekly sessions of 45 minutes. Patients in both conditions trained in groups of up to 8, supervised by a single person. The CRT and CC groups were scheduled at different times. The same personnel supervised both treatment conditions. All supervisors were trained by the coordinator of the study in the technical management of the two conditions.
  Other Names: Computerized active condition (CC)
  Arms: Computerized active condition
Other: Treatment as usual (TAU) — TAU: Patients in this condition participated in their (individually variable) daily rehabilitative activities. Patients allocated to the other two conditions also participated in these activities.
  Arms: Treatment as usual

SUMMARY:
Schizophrenia is known to be associated with cognitive dysfunction which increasing evidence suggests has consequences for functional adaptation and which cause difficulties in social re-integration after hospitalization. The investigators propose a large scale, multicentric study (7 centres from the Hermanas Hospitalarias del Sagrado Corazón de Jesús network) aimed at answering outstanding questions concerning the effectiveness of cognitive estimulation therapy for schizophrenic cognitive impairment. Specifically, the study will examine a) issues related to the size of the effect compared to treatment as usual and compared to a control intervention; b) generalizability of improvement to cognitive function and social cognition in daily life; and c) the durability of therapeutic gains after the end of treatment. 192 patients with chronic schizophrenia will be randomly assigned to one of three treatment conditions: a computer- assisted cognitive estimulation program (n=64), non-structured time on computer (n=64) and treatment as usual (n=64). A battery of neurocognitive tests of memory and executive function, including 'ecologically valid' measures, will be administered by blind evaluators at baseline, after 6 months of cognitive estimulation, and after 6 months follow-up. Symptoms, social functioning and self-esteem will be also be assessed at baseline, after the treatment and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or schizoaffective disorder fulfilling the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria diagnosis
* estimated premorbid intelligence quotient (IQ) in the normal range
* chronic illness (i.e. duration ≥two years)
* relative clinical stability (i.e. the patients had not experienced any recent exacerbation of symptoms).

Exclusion Criteria:

* history of brain trauma
* alcohol or substance abuse/dependence within the previous six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Memory test battery | Six months
  memory test battery Rivermead Behavioural Memory Test (RBMT)(Wilson, 1985) a memory test battery and the executive test battery, the Behavioural Assessment of the Dysexecutive Syndrome (BADS)(Wilson, 1996)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J McKenna, MD, Study Director — FIDMAG Germanes Hospitalàries Research Foundation; Jesus J Gomar, PhD, Principal Investigator — FIDMAG Germanes Hospitalàries Research Foundation; Edith Pomarol-Clotet, MD, PhD, Study Chair — FIDMAG Germanes Hospitalàries Research Foundation
Locations (1):
- FIDMAG Germanes Hospitalàries Research Foundation, Barcelona, Barcelona, Spain